CLINICAL TRIAL: NCT04941183
Title: A Randomized, Placebo-controlled, Double-blind, Single-ascending-dose and Multiple-ascending-dose, Phase 1 Study to Assess the Safety and Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of IV NTR-441 Solution in HV Adults and COVID-19 Patients
Brief Title: Phase 1 Study to Assess Safety, Tolerability, PD, PK, Immunogenicity of IV NTR-441 Solution in Healthy Volunteers and COVID-19 Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: the emergence of the omicron variant of COVID-19 lead to insufficient enrollment
Sponsor: Neutrolis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: NTR441-1001
Record Dates: First submitted 2021-05-04; First posted 2021-06-28 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Covid19
Keywords: Covid 19
MeSH Terms: conditions — COVID-19 | interventions — NTR-441

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, double-blind, single-ascending-dose and multiple-ascending-dose
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NTR-441 (Experimental): Single Ascending Dose; Multiple Ascending Dose.
  Interventions: Drug: NTR-441
- Placebo (Placebo Comparator): Single Ascending Dose; Multiple Ascending Dose.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NTR-441 — NTR-441
  Arms: NTR-441
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This first-in-human clinical study is a Phase 1a/ 1b, randomized, double-blind, placebo-controlled study to assess the safety, tolerability, and PK/PD of NTR-441 in healthy subjects and patients with COVID-19 after single ascending IV infusion doses and multiple ascending IV infusion doses.

ELIGIBILITY:
Healthy volunteers:

Inclusion Criteria:

* Male or female, non-smoker, ≥18 and ≤55 years of age, with Body Mass Index (BMI) > 18.5 and < 32.0 kg/m2
* Healthy with no clinically significant findings, determined by medical evaluation (medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory evaluations) at Screening
* Subject is able to understand and is willing to comply with all study requirements, and willing to follow the instructions of the study staff.
* Subject voluntarily agrees to participate in this study.

Exclusion Criteria:

* Pregnancy, nursing, and/or breastfeeding.
* Study participant has a history of an anaphylactic reaction.
* Subject has used an investigational drug within 30 days (or 5 half-lives whichever is longer) prior to the first dose of study drug.
* Has received any prescription or nonprescription over-the-counter (except occasional use of acetaminophen, paracetamol or ibuprofen) medication, topical medications, vitamins, dietary or herbal during the last 14 days or 5 half-lives, whichever is longer.
* Subject has a positive urine test for drugs of abuse at the screening visit or admission.
* Regular consumption of alcohol within 6 months prior to Screening or use of illicit substances within 3 months prior to screening.
* Subject has positive test for SARS-CoV-2 infection, human immunodeficiency virus (HIV), chronic or active hepatitis B, or active hepatitis C.
* Donation or loss of blood or plasma within 4 weeks prior to initial dosing.
* Subject has a history or current evidence of a serious and/or unstable cardiovascular, respiratory, gastrointestinal, hematologic, autoimmune, mental or other medical disorder, including cirrhosis or malignancy; a history of a psychiatric disorder that will affect the subject's ability to participate in the study.
* Subject has a clinically relevant abnormal ECG; abnormal laboratory values.
* Subject has hypertension.

COVID-19 patients:

Inclusion Criteria:

* Male or female, non-smoker, ≥18 years of age.
* Participant has active laboratory-confirmed SARS-CoV-2 infection.
* Participant must be hospitalized for COVID-19 pneumonia.
* Ability to provide informed consent personally, or by a legally acceptable representative if the participant is unable to do so.

Exclusion Criteria:

* Pregnancy, nursing, and/or breastfeeding.
* History of an anaphylactic reaction.
* In the opinion of the clinical team, progression to death is imminent and inevitable within the next 24 hours, irrespective of the provision of treatments.
* Severely immune-compromised participants.
* Participant known to test positive for human immunodeficiency virus (HIV), chronic or active hepatitis B, or active hepatitis C.
* Any other clinical conditions that in the opinion of the Investigator would make the participants unsuitable for the study.
* Prior treatment with any investigational drug therapy against coronavirus infection within 5 half-lives, prior to enrollment
* Participants who have received an experimental (or, in future, potentially a licensed) immunization or remdesivir against coronavirus remain eligible.
* Participation in another clinical study with the study intervention administered from 30 days or 5 half-lives whichever is longer.
* Anticipated transfer to another hospital which is not a study site during the intervention period.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
To evaluate safety and tolerability of single and multiple ascending doses of NTR-441 solution administered intravenously (IV) to adults | 60 days
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 following a single or multiple IV of NTR-441.

SECONDARY OUTCOMES:
Measurement of maximum plasma concentration (Cmax) | 15 days
  Maximum plasma concentration
Measurement of time of maximum plasma concentration (Tmax) | 14 days
  Time of maximum plasma concentration
Measurement of area under the concentration-time curve | 15 days
  Area under the concentration-time curve from predose to the time of the last quantifiable concentration
Measurement of the terminal elimination rate (λz) | 15 days
  Terminal elimination rate
Measurement of terminal elimination half-life (t½) | 15 days
  Terminal elimination half-life
Measurement of total body clearance (CL/F) | 15 days
  Total body clearance
Measurement of apparent volume of distribution | 15 days
  Apparent volume of distribution
To assess for immunogenicity of NTR-441 following single ascending and multiples ascending doses of NTR-441 solution administered IV to adults | 30 days
  Concentration of anti-drug antibodies of NTR-441 following single and multiples doses of NTR-441 solution administered IV

CONTACTS AND LOCATIONS:
Locations (4):
- Austria (2):
  - Klinik Favoriten, Vienna
  - Medical University Vienna, Department of Clinical Pharmacology, Vienna
- Ukraine (2):
  - Kyiv City Clinical Hospital#1, Kyiv
  - Vinnytsa City Clinical Hospital # 1, Vinnytsia

IPD SHARING:
Plan to Share IPD: No